CLINICAL TRIAL: NCT05293678
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Regeneron Anti-SARS-CoV-2 Monoclonal Antibody/Ies in Adult Healthy Volunteers
Brief Title: Safety and Tolerability of Regeneron Anti-SARS-CoV-2 Monoclonal Antibody/Ies in Adult Healthy Volunteers as Related to COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R15160-HV-2203; 2022-000182-41 (EudraCT Number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-24 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Vaccinated; Negative SARS-CoV2 Test Result
MeSH Terms: interventions — REGN15160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Lower IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (IV); Drug: Matching Placebo (IV)
- Mid IV Dose 1 (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (IV); Drug: Matching Placebo (IV)
- Mid IV Dose 2 (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (IV); Drug: Matching Placebo (IV)
- Higher IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (IV); Drug: Matching Placebo (IV)
- Lower SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (SC); Drug: Matching Placebo (SC)
- Mid SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (SC); Drug: Matching Placebo (SC)
- Higher SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN15160 (SC); Drug: Matching Placebo (SC)

INTERVENTIONS:
Drug: REGN15160 (IV) — Administered in single intravenous (IV) dose
  Arms: Higher IV Dose; Lower IV Dose; Mid IV Dose 1; Mid IV Dose 2
Drug: Matching Placebo (IV) — Administered in single IV dose
  Arms: Higher IV Dose; Lower IV Dose; Mid IV Dose 1; Mid IV Dose 2
Drug: REGN15160 (SC) — Administered in single subcutaneous (SC) dose
  Arms: Higher SC Dose; Lower SC Dose; Mid SC Dose
Drug: Matching Placebo (SC) — Administered in single SC dose
  Arms: Higher SC Dose; Lower SC Dose; Mid SC Dose

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of REGN15160 in healthy participants, as measured by all treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs).

The secondary objectives of the study are:

* To assess the concentration-time profile of REGN15160 in serum
* To assess the immunogenicity of REGN15160

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a SARS-CoV-2 negative test result from a sample collected ≤72 hours prior to randomization using a local reverse transcription polymerase chain reaction (RT-PCR) test or other molecular diagnostic assay and sample collection following assay standards
2. Has received complete primary series of standard-of-care COVID-19 vaccination per local guidance, completed at least 2 weeks prior to screening
3. Has a body mass index (BMI) between 18 and 31 kg/m2 (inclusive) at the screening visit
4. Is judged by the investigator to be in good health based on medical history, as defined in the protocol
5. Is in good health based on laboratory safety testing obtained at the screening visit

Key Exclusion Criteria:

1. History of clinically significant disease and any concern, as defined in the protocol and as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation
2. Was hospitalized (ie, >24 hours) for any reason within 30 days of the screening visit
3. Has history of alcohol or drug abuse as determined by the investigator
4. Has a history of significant multiple and/or severe allergies (eg, latex gloves), or has had an anaphylactic reaction to prescription or non-prescription drugs or food
5. Use of any prescription and non-prescription medications or nutritional supplements within approximately 5 half-lives or 2 weeks, whichever is longer, prior to first administration of the study drug through the end of the study, except for the permitted medications listed
6. Participated in any clinical research study evaluating another investigational drug including biologics or therapy, including specific immunotherapy, within at least 5 half-lives or 90 days (whichever is longer) of an investigational biologic drug, or at least 4 weeks for small molecules or other investigational drugs, prior to the screening visit
7. Is a pregnant or breastfeeding woman
8. Is a woman of childbearing potential (WOCBP)1 who is unwilling to practice highly effective contraception (as defined in the protocol) prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after study drug administration

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Occurrence and severity of all treatment emergent adverse events (TEAEs) | Through Day 169
Occurrence and severity of all serious adverse events (SAEs) | Through Day 169

SECONDARY OUTCOMES:
Concentrations of REGN15160 in serum | Through Day 169
Incidence and titer of anti-drug antibodies (ADA) to REGN15160 | Through Day 169

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Study Site, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/